CLINICAL TRIAL: NCT01928849
Title: Regional Anesthesia and Valproate Sodium for the Prevention of Chronic Post-Amputation Pain
Brief Title: Valproic Acid for the Prevention of Post-Amputation Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00047194; PT110575 (Other Grant/Funding Number: US Department of Defense)
Record Dates: First submitted 2013-02-15; First posted 2013-08-27 (Estimated); Results first posted 2018-10-25 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Pain, Phantom; Pain, Neuropathic
Keywords: Amputation; Post-amputation Pain; Neuropathic pain; Valproic Acid; Anesthesia, Conduction; Neuralgia, stump
MeSH Terms: conditions — Phantom Limb; Neuralgia | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cherry syrup (Placebo Comparator): Cherry Syrup: Patients randomized to the "Control arm" of the trial will receive standard regional anesthesia catheters (either peripheral nerve or epidural catheter), anesthetic management and the placebo.
  Interventions: Other: Cherry Syrup
- Valproic Acid (Experimental): "Intervention arm" patients will receive standard regional anesthesia catheters (either peripheral nerve or epidural catheter), anesthetic management, and valproic acid.
  Interventions: Drug: Valproic Acid

INTERVENTIONS:
Drug: Valproic Acid — "Intervention" patients will receive standard regional anesthesia catheters (either peripheral nerve or epidural catheter), anesthetic management and oral valproic acid 250mg preoperatively, then three times per day for either 6 days post-operatively or until discharge from the hospital.
  Other Names: Depacon, Depakene, Depakote, Stavzor
  Arms: Valproic Acid
Other: Cherry Syrup — Intervention arm patients will receive standard regional anesthesia catheters (either peripheral nerve or epidural catheter), anesthetic management, and valproic acid 250mg preoperatively, and then three times per day for 6 days post-operatively.
  Arms: Cherry syrup

SUMMARY:
The objectives of this study are, to test the effectiveness of Valproic Acid (VPA) in the prevention of chronic neuropathic and post-amputation pain, as well as to further define the underlying inflammatory and epigenetic mechanisms that lead to the development of such chronic pain.

HYPOTHESES AND QUESTIONS

Hypothesis 1: The use of oral valproic acid in combination with regional anesthesia in surgical limb-injury patients will decrease the incidence of chronic nerve injury and post-amputation pain.

Goal 1: In a blinded, randomized placebo-controlled, multi-center clinical trial, investigators will determine if oral VPA added to regional anesthesia and standard perioperative management will reduce the incidence of nerve injury and post-amputation pain when compared with regional anesthesia alone.

Hypothesis 2: The transition from acute to chronic pain is mediated via epigenetic mechanisms (differential DNA methylation) in genes involved in nociception.

Goal 2: Investigators will analyze the DNA methylation patterns of patients with different types of neuropathic and post-amputation pain and determine if they are altered by VPA.

DETAILED DESCRIPTION:
RESEARCH DESIGN

This study will be a prospective, randomized, double-blinded, placebo-controlled trial to test the efficacy of valproic acid (VPA) in reducing the incidence of chronic neuropathic and post-amputation pain following amputation, stump revision, and surgery for limb injury with neurologic damage. Patients randomized to the "Control arm" of the trial, will receive standard regional anesthesia catheters (either peripheral nerve or epidural catheter), anesthetic management and a placebo. Patients randomized to the "Intervention arm" of the trial will receive standard regional anesthesia catheters (either peripheral nerve or epidural catheter), anesthetic management, and valproic acid 250mg preoperatively, and then three times per day for either 6 days post-operatively or until the time of discharge.

METHODOLOGY

The enrollment goal for the study (from all sites) will be 224 patients. Subjects will be recruited from the surgical clinics and the anesthesia pre-operative clinic. Outcomes for patients in the intervention arm will be compared with those managed with the current institutional standards of care including regional anesthesia catheter infusions. The study team anticipates a 10% drop-out rate at 3 months secondary to death and loss to follow up. Thus 202 evaluable patients (101 patients in each arm) at 3 months after surgery will be included in this study.

After screening and enrollment, the study medication (VPA or placebo) will be administered. Research blood samples will be collected preoperatively, postoperatively (at the completion of study drug administration, and at the Amputation Clinic follow-up for expression analysis. The third and final blood draw will be taken at the 3 month follow up. If patient is unavailable the research team will make accommodations to collect blood sample at the 6 month follow up or at a time of maximal patient convenience, not to exceed 18 months from study enrollment. All samples will be de-identified and subsequently studied in our laboratory and core facilities at Duke. Study specific questionnaires will be administered during the hospital stay, at 1 month (via mail), at 3 months (in clinic) and at 6 months (in clinic when possible).

RANDOMIZATION AND TREATMENT

Randomization will be stratified by site and by surgical etiology. At the time of enrollment, subjects will be assigned to one of three surgical categories on the randomization assignment log: amputation, stump revision, or surgery for limb injury with neurologic damage. Prior to surgery, the Investigational Drug Pharmacist will dispense the study medication in liquid form and the container will be labeled "study drug" with no indication of the liquid contents. The pharmacist will be the only person aware of the treatment allocation. At the end of the trial, once endpoint adjudication has been completed for all study subjects, the study data and treatment allocation will be un-blinded. Initial drug administration will be performed prior to induction of anesthesia on the day of surgery. Subsequent doses will be administered at the bedside by the ICU or floor nurse depending on patient location. Participants will complete study drug administration unless they withdraw their consent or either their treating physician or the principal investigator believes it would be dangerous to continue valproic acid. If the subject withdraws during the administration of VPA, they will continue with their current medical regimen without alteration.

DATA ANALYSIS PLAN

The primary endpoint is the incidence of chronic pain at the 3 months or time of final adjudication evaluation point, and the chronic pain will be defined as an S-LANSS average pain score of 3 points or greater. Secondary endpoints will include the numeric scores from forms BPI, S-LANSS, and DVPRS and the change in these scores from baseline to 3 months or time of final adjudication, as well as the incidence of neuropathic limb or post-amputation pain at enrollment and 3 months or time of final adjudication. Frequency and percentage of the categorical variables in above endpoints will be reported by treatment arm and by assessed time. Mean, standard deviation and range of the mean scales of the above forms, as well as the changes of mean scales from baseline will be computed by arm and by assessed time. Two-sample chi-square tests will be used to assess the treatment difference of the primary endpoint and post-amputation pain (or neuropathic pain) at each time. Logistic regression will be applied to investigate the treatment difference on the primary endpoint and post-amputation pain by adjusting for potential prognostic variables including baseline pain level, study site, type of surgery, diabetes, and intervening therapies. Similar analyses will be carried out in study sub-groups of site, surgery type, and diabetic status. Two sample t-tests will be used to assess treatment difference in changes of mean scales from baseline. In addition, linear regression will be used to assess the treatment difference on changes of mean scales from baseline by adjusting for covariants. P values of less than 0.05 will be considered to indicate statistical significance. Intent-to-treat analysis will be performed. Sensitivity analyses will also be carried out by excluding patients who drop out before 3 month post-surgery. If the dropout rate is larger than 10% and if there is evidence that the missing mechanism is not MCAR (missing completely at random) but MAR (missing at random), multiple imputation will be conducted. RASS will be used during hospitalization to define any changes in sedation between study groups during drug administration.

Analysis of clinical study data will be carried out with a de-identified download from REDCap. All of these data shared with the Duke Center for Human Genetics (CHG) will be fully stripped of all 18 Health Insurance Portability and Accountability Act (HIPAA)identifiers (ID). Private health information of study participants will be respected and all data analysis will be done in blinded fashion, such that individuals will not be identifiable from the final analysis dataset. Each patient will be allocated a study ID number when they sign a consent form, and thereafter will be referred to by that number. Investigators will have secure password protected access to REDCap in order to enter data. The dataset and biorepository will be fully de-identified once the dataset is complete and locked.

Research blood samples are tracked and stored within our existing Laboratory Inventory Management System. All specimens are identified by barcode and are not identifiable except via a coding table held securely at Duke University Medical Center (DUMC), Durham Veterans Administration Medical Center (VAMC) and Walter Reed National Military Medical Center (WRNMMC) respectively.

ELIGIBILITY:
Inclusion Criteria:

* Male and female active duty military personnel or veterans, age 18 years and older.
* Patient is scheduled to undergo amputation, stump revision, or surgery for a limb injury with neurologic damage.
* Patient able to provide written informed consent prior to any study procedures.

Exclusion Criteria:

* Severe Traumatic Brain Injury (Diagnosis of traumatic brain injury resulting in documented, permanent or prolonged cognitive deficits that would preclude participation in the study)
* Significant cognitive deficits or dementia of any cause as noted in Computerized Patient Record System(CPRS).
* Patient has a designated Legally Authorized Representative
* Substantial hearing loss without alternative means of communication.
* Patient has documented spinal cord injury with permanent or persistent deficits
* Patient is under age 18 or a legal Minor
* Current pregnancy or lactation
* Cirrhosis with evidence of decompensation: coagulopathy International Normalized Ratio (INR) >1.3, thrombocytopenia with platelets <100,000, ascites or hepatic encephalopathy
* Therapy with valproic acid or other valproates, coumadin, chlorpromazine and olanzapine at the time of surgery and study drug administration
* Current diagnosis of seizure disorder requiring anti-epileptic medication
* Current therapy with tricyclic antidepressants (eg: amitriptyline, nortriptyline, imipramine, desipramine) at doses greater than 50mg/day
* Currently taking zidovudine
* Current diagnosis of malaria requiring anti-malaria medication (such as mefloquine and chloroquine)
* Currently taking monoamine oxide inhibitors (MAOI)
* Allergy to valproates or valproic acid
* Contraindication to, or refusal of, regional anesthesia catheter
* BMI > 50

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2013-12; Primary Completion 2017-09-26 (Actual); Study Completion 2017-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Buchheit, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Duham VA Medical Center, Durham, North Carolina

REFERENCES:
- [Background] Gill D, Derry S, Wiffen PJ, Moore RA. Valproic acid and sodium valproate for neuropathic pain and fibromyalgia in adults. Cochrane Database Syst Rev. 2011 Oct 5;2011(10):CD009183. doi: 10.1002/14651858.CD009183.pub2. PMID 21975791
- [Background] Sinn DI, Kim SJ, Chu K, Jung KH, Lee ST, Song EC, Kim JM, Park DK, Kun Lee S, Kim M, Roh JK. Valproic acid-mediated neuroprotection in intracerebral hemorrhage via histone deacetylase inhibition and transcriptional activation. Neurobiol Dis. 2007 May;26(2):464-72. doi: 10.1016/j.nbd.2007.02.006. Epub 2007 Feb 23. PMID 17398106
- [Background] Detich N, Bovenzi V, Szyf M. Valproate induces replication-independent active DNA demethylation. J Biol Chem. 2003 Jul 25;278(30):27586-92. doi: 10.1074/jbc.M303740200. Epub 2003 May 14. PMID 12748177
- [Background] Zhang Z, Cai YQ, Zou F, Bie B, Pan ZZ. Epigenetic suppression of GAD65 expression mediates persistent pain. Nat Med. 2011 Oct 9;17(11):1448-55. doi: 10.1038/nm.2442. PMID 21983856
- [Background] Reiber GE, McFarland LV, Hubbard S, Maynard C, Blough DK, Gambel JM, Smith DG. Servicemembers and veterans with major traumatic limb loss from Vietnam war and OIF/OEF conflicts: survey methods, participants, and summary findings. J Rehabil Res Dev. 2010;47(4):275-97. doi: 10.1682/jrrd.2010.01.0009. PMID 20803399

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cherry Syrup | Valproic Acid
Started | 66 | 62
Completed | 52 | 55
Not Completed | 14 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cherry Syrup | Valproic Acid | Total
Number analyzed (Participants) | 66 | 62 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (16.6) | 51.1 (18.2) | 50.7 (17.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 55 | 51 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 63 | 59 | 122
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 12 | 27
  White | 49 | 49 | 98
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 66 | 62 | 128

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Chronic Post-amputation Pain
Description: The primary endpoint is the incidence of chronic pain after surgery. The study team will use the average pain score over the past week as noted on the Self-Reported Leeds Assessment of Neuropathic Symptoms and Signs pain scale (S-LANSS) for the assessment of pain, and define chronic pain as a score greater than or equal to 3.
Time Frame: 3 months or time of final adjudication assessment, up to 6 months
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cherry Syrup | Valproic Acid
Number analyzed (Participants) | 52 | 55
Participants | 37 | 36
Statistical Analysis 1: Comparison: Cherry Syrup vs Valproic Acid; Test type: Other; p = 0.53, Regression, Logistic; Univariable Logistic regression; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.34 to 1.74]

2. Secondary Outcome: Incidence of Pain Sub-types
Description: The incidence of neuropathic limb or post-amputation pain sub-types as defined by adjudication classification at each assessment time point.
Time Frame: Assessments at enrollment and 3 months or time of final adjudication assessment (up to 6 months)
Population: Participants who completed the study. For the cherry syrup (placebo) arm, only 50 participants completed the full adjudication process necessary to determine phantom pain sub-type.
Measure: Count of Participants; unit: Participants
Arm/Group | Cherry Syrup | Valproic Acid
Number analyzed (Participants) | 52 | 55
Participants
  Residual limb pain | 29 | 31
  Phantom limb: number analyzed (Participants) | 50 | 55
  Phantom limb | 22 | 26
Statistical Analysis 1: Comparison: Cherry Syrup vs Valproic Acid; Comparison of rate of residual limb pain between treatment groups; Test type: Other; p = 0.95, Chi-squared
Statistical Analysis 2: Comparison: Cherry Syrup vs Valproic Acid; Comparison of rate of Phantom limb pain between treatment groups; Test type: Other; p = 0.74, Chi-squared

3. Secondary Outcome: Effect on Analgesic Requirement
Description: The effect of study drug on perioperative analgesic consumption and corresponding analysis of pain/sedation scales. Outcome defined as total opioid consumption (mg) during each 24-hour periods following surgery.
Time Frame: Assessments during hospitalization (0-24 hours and 24-48 hours post-surgery)
Population: Patients who completed the study
Measure: Median (Inter-Quartile Range); unit: morphine milligram equivalents
Arm/Group | Cherry Syrup | Valproic Acid
Number analyzed (Participants) | 52 | 55
morphine milligram equivalents
  Postoperative hours 0-24 | 59 [20 to 89] | 33 [20 to 114]
  Postoperative hours 24-48 | 49 [24 to 159] | 45 [20 to 114]
Statistical Analysis 1: Comparison: Cherry Syrup vs Valproic Acid; Comparison of opioid consumption postoperative hours 0-24; Test type: Other; p = 0.27, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cherry Syrup vs Valproic Acid; Comparison of opioid consumption postoperative hours 24-48; Test type: Other; p = 0.27, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Brief Pain Inventory (BPI) Short Form Score
Description: The BPI short form is a multidimensional patient-completed measure that assesses the sensory component of pain intensity. We will analyze the change in average pain score question (ranges 0-10) and the sum of the 7 interference questions (total range 0-70) from baseline. Higher score indicates greater pain and interference.
Time Frame: Assessments at enrollment and 3 months or time of final adjudication assessment (up to 6 months)
Population: Those completing questionnaires at both time points
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cherry Syrup | Valproic Acid
Number analyzed (Participants) | 49 | 53
score on a scale
  BPI Average Pain Score: number analyzed (Participants) | 49 | 52
  BPI Average Pain Score | -2 [-3 to 0] | -1 [-3 to 0]
  BPI interference question sum | -15 [-33 to -4] | -7 [-31 to 0]
Statistical Analysis 1: Comparison: Cherry Syrup vs Valproic Acid; Comparison of BPI average pain score; Test type: Other; p = 0.59, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cherry Syrup vs Valproic Acid; Comparison of BPI Interference question sum; Test type: Other; p = 0.16, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Self-Reported Leeds Assessment of Neuropathic Symptoms and Signs Pain Scale (S-LANSS)
Description: The S-LANSS is a self-reported version of the Leeds Assessment of Neuropathic Symptoms and Signs pain scale. It aims to differentiate neuropathic pain from somatic or nociceptive pain. We will analyze the change in numeric average pain score during the past week (range from 0-10) from baseline. Higher scores indicate greater pain.
Time Frame: Assessments at enrollment and 3 months or time of final adjudication assessment (up to 6 months)
Population: Patients who completed questionnaire at both time points
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cherry Syrup | Valproic Acid
Number analyzed (Participants) | 52 | 55
score on a scale | -2 [-5 to -1] | -2 [-5 to 0]
Statistical Analysis 1: Comparison: Cherry Syrup vs Valproic Acid; Test type: Other; p = 0.35, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Defense and Veterans Pain Rating Scale (DVPRS) Score
Description: The DVPRS is a pain assessment tool developed by the military in an effort to improve reliability and interpretability of pain assessment in the military population. It has been found to be an effective and valid tool in this population. We will analyze the change in numeric pain response (range 0-10) and the sum of the four supplemental questions (range 0-40) from baseline. Higher scores indicate greater pain and functional limitations.
Time Frame: Assessments at enrollment and 3 months or time of final adjudication assessment (up to 6 months)
Population: Patients who completed questionnaires at both time points
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cherry Syrup | Valproic Acid
Number analyzed (Participants) | 43 | 46
score on a scale
  DVPRS numeric pain: number analyzed (Participants) | 43 | 44
  DVPRS numeric pain | -2 [-3 to 0] | 0 [-3.5 to 0]
  DVPRS Supplemental Question Sum | -9 [-18 to -1] | -4.5 [-17 to 0]
Statistical Analysis 1: Comparison: Cherry Syrup vs Valproic Acid; Comparison of DVPRS numeric pain score; Test type: Other; p = 0.42, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cherry Syrup vs Valproic Acid; Comparison of DVPRS supplemental question sum; Test type: Other; p = 0.19, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Richmond Agitation-Sedation Scale (RASS)
Description: The RASS is a commonly used, valid and reliable assessment tool for use in hospitalized patients. Validity testing reveals good inter-rater reliability among medical, surgical, and intensive care units. We will analyze the numeric score at each assessment (range -5 (unarousable) to 4 (combative)).
Time Frame: during hospitalization (0-24 hours and 24-48 hours post-surgery)
Population: Participants who completed the RASS assessment on post-op day 1.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cherry Syrup | Valproic Acid
Number analyzed (Participants) | 47 | 51
score on a scale
  Post-op hours 0-24: number analyzed (Participants) | 47 | 50
  Post-op hours 0-24 | 0 [0 to 0] | 0 [0 to 0]
  Post-op hours 24-48: number analyzed (Participants) | 45 | 51
  Post-op hours 24-48 | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Cherry Syrup vs Valproic Acid; Comparison of RASS postoperative hours 0-24; Test type: Other; p = 0.27, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cherry Syrup vs Valproic Acid; Comparison of RASS postoperative hours 24-48; Test type: Other; p = 0.26, Wilcoxon (Mann-Whitney)

8. Other Pre Specified Outcome: Observation of Epigenetic Alterations That Occur in the Transition From Acute to Chronic Pain.
Description: Epigenetic analysis (DNA methylation) will be correlated with pain sub-type and use of Valproic Acid.
Time Frame: Changes between enrollment, end of study drug and 3 months or time of final adjudication
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Severe adverse events were collected from surgery to 3 months or time of final adjudication assessment (up to 6 months)
Arm/Group | Cherry Syrup | Valproic Acid
All-Cause Mortality (participants affected / at risk) | 4/66 | 2/62
Serious Adverse Events (participants affected / at risk) | 26/66 | 20/62
Other Adverse Events (participants affected / at risk) | 31/66 | 27/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cherry Syrup (N=66) | Valproic Acid (N=62)
Cardiac Disorders (Cardiac disorders) | 1 (1) | 2 (2)
Blood and lymphatic system disorder (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Endocrine disorder (Endocrine disorders) | 1 (1) | 0 (0)
Gastrointestinal discorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vascular Disorder (Vascular disorders) | 0 (0) | 1 (1)
Infections and infestations (Infections and infestations) | 7 (7) | 4 (4)
Nervous system disorders (Nervous system disorders) | 3 (3) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Surgical and medical procedures (Surgical and medical procedures) | 7 (7) | 8 (8)
General Disorder (General disorders) | 7 (7) | 2 (2)
Renal and urinary disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cherry Syrup (N=66) | Valproic Acid (N=62)
Hepatobiliary disorder (Hepatobiliary disorders) | 7 (7) | 4 (4)
Gastrointestinal disorder (Gastrointestinal disorders) | 4 (4) | 10 (10)
Infection and infestations (Infections and infestations) | 9 (9) | 8 (8)
Nervous System disorder (Nervous system disorders) | 5 (5) | 3 (3)
Injury, poisoning and procedural complication (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Surgical and medical procedures (Surgical and medical procedures) | 6 (6) | 3 (3)
General Disorders (General disorders) | 7 (7) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT01928849/Prot_SAP_000.pdf